CLINICAL TRIAL: NCT06976866
Title: Effect of Topical Application of Atorvastatin Gel Versus Hyaluronic Acid on Immediate Loading Dental Implant in Posterior Maxilla
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amira attia (Other)
Responsible Party: Sponsor-Investigator, Amira attia, assistant professor, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: M0103023OS
Record Dates: First submitted 2025-04-22; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: In Recent Years, There Has Been a Rise in the Use of Immediate Loading Protocols; Dental Implant Stability
Keywords: Immediate loading; Hyaluronic acid; Atorvastatin; ; Bone density; Posterior maxilla.

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- hyaluronic acid (Experimental): [Hyaluronic acid (HA) group]: 7 patients received implants coated with HA gel .
  Interventions: Procedure: implant surgery
- atorvastatin (Experimental): [atorvastatin (ATV) group]: 7 patients received implants coated with ATV gel
  Interventions: Procedure: implant surgery
- control (Experimental): group I (control group): 7 patients received implants without coating by any materials.
  Interventions: Procedure: implant surgery

INTERVENTIONS:
Procedure: implant surgery — surgery
  Other Names: hyaluronic acid around implant; atorvastatin around implant

SUMMARY:
Background: In recent years, there has been a rise in the use of immediate loading protocols; however, the complex anatomy of the posterior maxilla presents challenges. Currently, there is a lack of comparative studies assessing the effects of hyaluronic acid and atorvastatin gel on enhancing bone density in this region in conjunction with immediate loading. This study aimed to compare the effect of topical application of atorvastatin gel versus hyaluronic acid around immediately loaded dental implant that replacing missed maxillary posterior teeth.

Patients and methods: twenty one patients were chosen from the Outpatient Clinic in the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University seeking implant placement. Patients were divided randomly and equally into three groups: group I (control group): 7 patients received implants without coating by any materials. Group II [Hyaluronic acid (HA) group]: 7 patients received implants coated with HA gel .Group III [atorvastatin (ATV) group]: 7 patients received implants coated with ATV gel. Clinical evaluation of implant stability was performed at the time of implant insertion and after 3 and 6 months postoperative. Also, peri-implant pocket depth (PPD) and modified sulcus bleeding index (mSBI) were evaluated. Radiographical evaluation of bone density (BD) was performed immediately and after 6 months postoperatively of implant loading using CBCT. All clinical and radiographic data were subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria:

* patients with one or more missing maxillary posterior teeth
* age ranging from 18 to 45 years
* patient's cooperation
* motivation and good oral hygiene
* adequate occlusion (proper interarch space).

Exclusion Criteria:

* individuals with systemic or local diseases that are contraindicative of surgery or implant placement
* pregnant individuals
* individuals with any bone diseases that may impede bone healing
* smokers
* individuals who exhibit parafunctional habits like bruxism and clenching.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-05-13 (Estimated); Study Completion 2025-05-14 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation | 6 months
  Clinical evaluation of implant stability was performed at the time of implant insertion and after 3 and 6 months postoperative.
clinical evaluation | 6 months
  Clinical evaluation of implant stability was performed at the time of implant insertion and after 3 and 6 months postoperative. Also, peri-implant pocket depth (PPD) and modified sulcus bleeding index (mSBI) were evaluated.
clinical evaluation | 6 months
  peri-implant pocket depth (PPD) around the implant at 3 months and 6 months after loading

SECONDARY OUTCOMES:
radiographic evaluation | 6 months
  Radiographical evaluation of bone density (BD) was performed immediately and after 6 months postoperatively of implant loading using CBCT
clinical evaluation | 6 months
  modified sulcus bleeding index (mSBI) were evaluated at 3 months and 6 months after loading

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Attia, Al Mansurah, Egypt